CLINICAL TRIAL: NCT02935257
Title: Immunotherapy for High Risk/Relapsed CD19+ Acute Lymphoblastic Leukaemia, B-cell Non-Hodgkin's Lymphoma (B-NHL) and Chronic Lymphocytic Leukaemia (CLL)/ Small Lymphocytic Lymphoma (SLL) Using CAR T-cells to Target CD19
Acronym: ALLCAR19
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/16/0530
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Lymphoblastic, Acute, Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19CAT-41BBZ CAR T-cells (Experimental): Treatment with the ATIMP: CD19CAT-41BBZ CAR T-cells
  Interventions: Biological: CD19CAT-41BBZ CAR T-cells

INTERVENTIONS:
Biological: CD19CAT-41BBZ CAR T-cells — Infusion with CD19CAT-41BBZ CAR T-cells

SUMMARY:
This is a multi-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) in adults (age ≥16) with (1) high risk, relapsed/refractory (r/r) CD19+ B-ALL; (2) r/r DLBCL; (3) r/r CLL/SLL and (4) r/r FL and (5) r/r MCL. The ATIMP for this study is cryopreserved autologous patient-derived T-cells transduced with the lentiviral pCCL.PGK.alpha.CD19CAT-41BBzeta vector, CD19CAT-41BBζ CAR T-cells (referred to subsequently as CD19CAR T-cells) which is classified as a gene therapy medicinal product. Patients will undergo an unstimulated leucapheresis for the generation of the ATIMP. The ATIMP will take approximately 15 days to generate. During this period, patients may receive "holding" chemotherapy as per institutional practice to maintain disease control. The study will evaluate ATIMP safety and efficacy and the duration of disease response in adults with high risk / relapsed CD19+ B-ALL, DLBCL, B-CLL/SLL, FL and MCL.

Recruitment into the ALL cohort has been completed and no further patients with ALL are being treated on the study.

Patients receive pre-conditioning lymphodepleting chemotherapy with cyclophosphamide 60mg/kg on Day -6 and fludarabine 30mg/m2 administered over 3 days (Day -5 to Day -3). Patients with DLBCL only will also receive a single dose of pembrolizumab 200 mg at day -1.

Patients recruited to ALLCAR19 are treated with different dosing schedules, depending on their underlying disease. Patients with B-ALL and B-CLL/SLL are considered at high risk of CLL/CRES so receive split dosing, with the second dose only given in the absence of severe toxicity 9 days later. CAR T-cell dosing in ALLCAR19 is flat i.e. not dependent on patient body weight or surface area.

* Regimen A1: Patients with B-ALL with a baseline marrow blast% of ≤20% receive a split dose with a first dose of 100 x 10^6 CD19 CAR T-cells and a possible second dose of 310 x 106 CAR T-cells
* Regimen A2: Patients with B-ALL with a baseline marrow blast% of >20% receive a split dose with a first dose of 10 x 10^6 CD19CAR T-cells and a possible second dose of 400 x 10^6 CAR T-cells
* Regimen B: Patients with DLBCL receive a single dose of 200 x 10^6 CAR T-cells
* Regimen C: Patients with CLL/SLL will receive a split dose with a first dose of 30 x 106 CD19 CAR T-cells and a possible second dose of 200 x 10^6 CD19 CAR T-cells.
* Regimen D: Patients with FL and MCL receive a single dose of 200 x 10^6 CAR T-cells

The study evaluates ATIMP feasibility and safety of generating CD19CAR T-cells and for B-ALL patients only, efficacy and the duration of disease response to CD19CAR T-cells.

After completing the interventional phase of the study all patients, irrespective of whether they progressed or responded to treatment, enter long term follow up until 10 years post-CD19CAR T-cell infusion.

DETAILED DESCRIPTION:
This is a multi-centre, non-randomised, open label Phase I clinical trial of an Advanced Therapy Investigational Medicinal Product (ATIMP) in adults (age ≥16) with (1) high risk, relapsed/refractory (r/r) CD19+ B-ALL; (2) r/r DLBCL; (3) r/r CLL/SLL, (4) r/r FL and (5) r/r MCL. The ATIMP for this study is cryopreserved autologous patient-derived T-cells transduced with the lentiviral pCCL.PGK.alpha.CD19CAT-41BBζ vector, CD19CAT-41BBζ CAR T-cells (referred to sub-sequently as CD19CAR T-cells) which is classified as a gene therapy medicinal product. Patients will undergo an unstimulated leucapheresis for the generation of the ATIMP. The ATIMP take approximately 15 days to generate. During this period, patients may receive "holding" chemotherapy as per institutional practice to maintain disease control. The study evaluates ATIMP safety and efficacy and the duration of disease response in adults with high risk / relapsed CD19+ B-ALL, DLBCL, B-CLL/SLL, FL and MCL.

The ALL and FL cohorts are now completed and no further patients with ALL or FL are treated on the study.

Patients receive lymphodepleting chemotherapy with cyclophosphamide 60mg/kg on Day -6 and fludarabine 30mg/m2 administered over 3 days (Day -5 to Day -3). Patients with DLBCL only also receive a single dose of pembrolizumab 200 mg at day -1.

Patients recruited to ALLCAR19 are treated with different dosing schedules, depending on their underlying disease. Patients with B-ALL and B-CLL/SLL are considered at high risk of CLL/CRES so receive split dosing, with the second dose only given in the absence of severe toxicity 9 days later. CAR T-cell dosing in ALLCAR19 is flat i.e. not dependent on patient body weight or surface area.

* Regimen A1: Patients with B-ALL with a baseline marrow blast% of ≤20% receive a split dose with a first dose of 100 x 10^6 CD19 CAR T-cells and a possible second dose of 310 x 10^6 CAR T-cells
* Regimen A2: Patients with B-ALL with a baseline marrow blast% of >20% receive a split dose with a first dose of 10 x 10^6 CD19CAR T-cells and a possible second dose of 400 x 106 CAR T-cells
* Regimen B: Patients with DLBCL receive a single dose of 200 x 10^6 CAR T-cells
* Regimen C: Patients with CLL/SLL will receive a split dose with a first dose of 30 x 10^6 CD19 CAR T-cells and a possible second dose of 200 x 106 CD19 CAR T-cells.
* Regimen D: Patients with indolent B-NHL receive a single dose of 200 x 10^6 CAR T-cells

The study evaluates ATIMP feasibility and safety of generating CD19CAR T-cells and for B-ALL patients only, efficacy and the duration of disease response to CD19CAR T-cells.

After completing the interventional phase of the study all patients, irrespective of whether they progressed or responded to treatment, will enter long term follow up until 10 years post-CD19CAR T-cell infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥162. B-ALL: high risk or relapsed histologically confirmed CD19+ B-ALL following standard therapy requiring salvage in whom alternative therapies are deemed inappropriate by their treating physician Or DLBCL: relapsed/refractory DLBCL (incl. transformed FL but not Richter's transformation) following ≥2 prior lines of therapy including Rituximab and anthracycline Or CLL/SLL: relapsed/refractory CLL/SLL following ≥2 prior lines of therapy including Ibrutinib or other Bruton's Tyrosine Kinase (BTK) inhibitors Or Follicular Lymphoma which is relapsed / refractory following ≥2 prior lines of therapy Or Mantle Cell Lymphoma which is relapsed / refractory following ≥2 prior lines of therapy 3. Agreement to have a pregnancy test, use adequate contraception (if applicable) 4.Written informed consent

Exclusion criteria for registration:

1. CD19 negative disease
2. B-ALL and CLL: overt CNS involvement (i.e.: patients with CNS2 with neurological symp-toms or patients with CNS3; appendix 2)
3. DLBCL, FL, MCL and CLL/SLL: primary or secondary CNS lymphoma
4. Isolated extramedullary disease (B-ALL and CLL)
5. Active hepatitis B, C or HIV infection
6. Oxygen saturation ≤ 90% on air
7. Bilirubin >2 x upper limit of normal
8. GFR <50ml/min
9. Women who are pregnant or breast feeding
10. Stem Cell Transplant patients only: active significant acute GVHD (overall Grade ≥ II, Seattle criteria) or moderate/severe chronic GVHD (NIH consensus criteria) requiring im-munosuppressive therapy and/or systemic steroids
11. Inability to tolerate leucapheresis
12. Karnofsky score <60% (see appendix 3)
13. Patients who have experienced significant neurotoxicity following blinatumomab
14. Known allergy to albumin or DMSO
15. Life expectancy <3months
16. Significant cardiac disease, left ventricular ejection fraction <40% and uncontrolled cardiac arrhythmias (patients with rate-controlled atrial fibrillation are not excluded)
17. Pre-existing neurological disorders (other than CNS involvement of underlying haemato-logical malignancy)
18. DLBCL only:

    * Any contraindications to PD-1 antibody Pembrolizumab
    * History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) re-sulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 24 months
    * Evidence of active pneumonitis on chest computed tomography (CT) scan at screening or history of drug-induced pneumonitis, idiopathic pulmonary fibrosis, organising pneu-monia (e.g. bronchiolitis obliterans), or idiopathic pneumonitis. Prior radiation pneu-monitis in the radiation field (fibrosis) is allowed (if >24 weeks since the event)
    * Chest/mediastinal radiation within 24 weeks of CAR T-cellinfusion

Exclusion criteria: for CD19CAR T-cell infusion at Day 0 (all patients):

1. Severe intercurrent infection at the time of scheduled CD19CAR T-cell infusion
2. Requirement for supplementary oxygen or active pulmonary infiltrates at the time of scheduled CD19CAR T-cell infusion
3. Allogeneic transplant recipients with active significant acute GVHD overall grade ≥II or moderate/severe chronic GVHD requiring systemic steroids or other immunosuppres-sion at the time of scheduled CD19CAR T-cell infusion. Note: Such patients will be ex-cluded until the patient is GVHD free and off steroids

Exclusion criteria: for supplementary CD19CAR T-cell infusion Day 9 (B-ALL and CLL/SLL patients):

1. Severe intercurrent infection at the time of scheduled CD19CAR T-cell infusion
2. Requirement for supplementary oxygen or active pulmonary infiltrates at the time of scheduled CD19CAR T-cell infusion
3. Grade 3-4 CRS and or grade 3-4 neurotoxicity following Day 0 CD19CAR T-cell dose
4. Grade 1-2 neurotoxicity (if occurred) following Day 0 CD19CAR T-cell dose that has not fully resolved prior to proposed administration of 2nd CD19CAR T-cell dose
5. Persisting Grade 2 CRS following Day 0 CD19CAR T-cell dose that has not resolved to ≤ Grade 1 CRS prior to proposed administration of 2nd CD19CAR T-cell dose
6. Allogeneic transplant recipients with active significant acute GVHD overall grade ≥II or moderate/severe chronic GVHD requiring systemic steroids or other immunosuppression at the time of scheduled CD19CAR T-cell infusion* *Note: Such patients will be excluded until the patient is GVHD free and off steroids

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity evaluated by the incidence of grade 3-5 toxicity causally related to the ATIMP | 28 days
  Toxicity following CD19CAR T-cell administration as evaluated by the incidence of grade 3-5 toxicity causally related to the ATIMP.
Feasibility of manufacturing CD19CAR T-cells evaluated by the number of therapeutic products generated | 30 days
  Feasibility of adequate leucapheresis collection and generation of CAR19 T cells as evaluated by the number of therapeutic products generated.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Peggs, Study Chair — University College London Hospitals
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roddie C, Dias J, O'Reilly MA, Abbasian M, Cadinanos-Garai A, Vispute K, Bosshard-Carter L, Mitsikakou M, Mehra V, Roddy H, Hartley JA, Spanswick V, Lowe H, Popova B, Clifton-Hadley L, Wheeler G, Olejnik J, Bloor A, Irvine D, Wood L, Marzolini MAV, Domning S, Farzaneh F, Lowdell MW, Linch DC, Pule MA, Peggs KS. Durable Responses and Low Toxicity After Fast Off-Rate CD19 Chimeric Antigen Receptor-T Therapy in Adults With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia. J Clin Oncol. 2021 Oct 20;39(30):3352-3363. doi: 10.1200/JCO.21.00917. Epub 2021 Aug 31. PMID 34464155